CLINICAL TRIAL: NCT03680144
Title: Diagnostic Accuracy of Dynamic Susceptibility Contrast (DSC) Perfusion MRI to Determine Radiation Necrosis Versus Tumor Progression in Brain Metastases Treated With Stereotactic Radiosurgery
Brief Title: Utility of Perfusion MRI to Detect Radiation Necrosis in Patients With Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Hui-Kuo Shu, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00102506; NCI-2018-01722 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD4391-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Invasive Malignant Neoplasm; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (MRI, DSC-MRI) (Experimental): Participants undergo diagnostic magnetic resonance imaging (MRI) with and without contrast and treatment planning dynamic susceptibility contrast-MRI (DSC-MRI) series before receiving SRS at 4-6 weeks after SRS, and then every 3 months unless clinically indicated sooner.
  Interventions: Procedure: Dynamic Susceptibility Contrast-MRI (DSC-MRI); Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Dynamic Susceptibility Contrast-MRI (DSC-MRI) — Undergo DSC-MRI
  Other Names: Dynamic Susceptibility Contrast-Enhanced MRI
Procedure: Magnetic Resonance Imaging (MRI) — Undergo diagnostic MRI
  Other Names: MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This trial studies how well dynamic susceptibility contrast-magnetic resonance imaging (MRI) works in determining radiation necrosis and tumor progression in participants with cancer that has spread to the brain and are being treated with radiation therapy. Diagnostic procedures, such as dynamic susceptibility contrast-MRI, may improve the ability to determine indeterminate post-treatment changes seen on imaging after radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To prospectively determine the sensitivity and specificity of dynamic susceptibility contrast (DSC)-MRI parameters in detecting tumor recurrence versus radiation necrosis for brain metastases treated with stereotactic radiosurgery (SRS).

SECONDARY OBJECTIVES:

I. To correlate radiographic diagnoses with pathologic diagnoses when surgical resection is clinically indicated.

II. To correlate baseline relative cerebral blood volume (rCBV) values and other hemodynamic parameters with tumor primary histology.

III. To assess overall survival, local failure, distant brain failure and neurologic death.

OUTLINE:

Participants undergo a diagnostic MRI with and without contrast and treatment planning DSC perfusion MRI series before receiving SRS at 4-6 weeks after SRS, and then every 3 months unless clinically indicated sooner.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of invasive malignancy with at least radiographic evidence of intracranial disease as seen on MRI.
* At least one identifiable intracranial lesion ≥ 1 cm in diameter enrolled within 4 weeks of diagnosis.
* Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2.

Exclusion Criteria:

* Planned whole-brain radiotherapy (WBRT) with boost.
* Leptomeningeal disease.
* Inadequate renal function (estimated glomerular filtration rate [eGFR] > 30 ml/min/1.73 m²) or contrast allergy.
* Non-MRI compatible pacemaker with pacemaker dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Change in dynamic susceptibility contrast (DSC)-magnetic resonance imaging (MRI) parameters: relative cerebral blood volume (rCBV) | Baseline up to 1 year
  Image processing will occur in a blinded manner using nordicICE software (NordicNeuroLab AS, Bergen, Norway). Signal-intensity curves will be created per voxel. Regions of interest will be designated around the contrast enhancing lesion as seen on T1-post contrast MR. An additional contralateral area of normal-appearing white matter will be designated in the same axial plane to standardize the data. rCBV is calculated as the ratio of the CBV within the enhancing region to the CBV within the contralateral normal-appearing white matter.
Change in dynamic susceptibility contrast (DSC)-magnetic resonance imaging (MRI) parameters: relative peak height (rPH) | Baseline up to 1 year
  Image processing will occur in a blinded manner using nordicICE software (NordicNeuroLab AS, Bergen, Norway). Signal-intensity curves will be created per voxel. Regions of interest will be designated around the contrast enhancing lesion as seen on T1-post contrast MR. An additional contralateral area of normal-appearing white matter will be designated in the same axial plane to standardize the data. rPH is defined as the maximal change in contrast signal intensity from pre-contrast baseline compared to the lowest signal intensity during contrast bolus, normalized to the signal in the contralateral normal-appearing white matter.
Change in dynamic susceptibility contrast (DSC)-magnetic resonance imaging (MRI) parameters: percentage of signal intensity recovery (PSR) | Baseline up to 1 year
  Image processing will occur in a blinded manner using nordicICE software (NordicNeuroLab AS, Bergen, Norway). Signal-intensity curves will be created per voxel. Regions of interest will be designated around the contrast enhancing lesion as seen on T1-post contrast MR. An additional contralateral area of normal-appearing white matter will be designated in the same axial plane to standardize the data. PSR is defined as the percentage of the difference between lowest signal intensity during contrast bolus and the recovery post-contrast signal intensity compared to the peak height.
Change in dynamic susceptibility contrast (DSC)-magnetic resonance imaging (MRI) parameters: mean transit time (MTT) | Baseline up to 1 year
  Image processing will occur in a blinded manner using nordicICE software (NordicNeuroLab AS, Bergen, Norway). Signal-intensity curves will be created per voxel. Regions of interest will be designated around the contrast enhancing lesion as seen on T1-post contrast MR. An additional contralateral area of normal-appearing white matter will be designated in the same axial plane to standardize the data. MTT is defined as the average time in which contrast passes through a given region of brain tissue and is estimated from the contrast concentration-time course curve (CC-TCC) as width of the curve at half maximum height.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Kuo Shu, MD, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

DOCUMENTS (1):
  • Informed Consent Form (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT03680144/ICF_000.pdf